CLINICAL TRIAL: NCT06172842
Title: Multi-modality Echocardiography for Cardiac Assessment in Primary Electrical Disease
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1069-01
Record Dates: First submitted 2023-11-24; First posted 2023-12-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Multi-modality Echocardiography; Primary Electrical Disease
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary electrical disease
  Interventions: Diagnostic Test: Echocardiography
- control
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Multi-modality echocardiography

SUMMARY:
From 2020 to 2023, patients with primary electrical disease (idiopathic ventricular fibrillation, long QT syndrome, Andersen-Tawil syndrome type I, Brugada syndrome, early repolarization syndrome, CPVT, and short QT syndrome) were first diagnosed at Sun Yat-sen Memorial Hospital of Sun Yat-sen University, and clinical data and echocardiographic indicators were recorded. Follow-up is until December 30, 2025 or endpoint event occurs. Endpoint events were defined as sustained ventricular tachycardia, ventricular fibrillation, sudden cardiac death, ICD discharge events, all-cause death, heart failure and heart transplantation, which were statistically analyzed as a composite endpoint of cardiovascular analysis. The predictors of primary electrical disease and the risk factors for adverse cardiovascular events were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* primary electrical disease

Exclusion Criteria:

* Congenital heart disease, poor echocardiographic images, moderate or severe valvular disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary electrical disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Multi-modality echocardiography | 2 years
  tissue Doppler imging, speckle-tracking-strain, myocardial work, mechanical dispersion,electro-mechanical window

CONTACTS AND LOCATIONS:
Locations (1):
- Hanlu Lv, Guangzhou, China